CLINICAL TRIAL: NCT05057286
Title: The Effect of a Combination Between Clinical Crown Lengthening Surgery and Botulinum Toxin A Injection in Gummy Smile Treatment
Brief Title: Effect of Clinical Crown Lengthening Surgery and Botulinum Toxin A Injection in Gummy Smile Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Thu Thuy, Deputy Head of Department of Periodontology, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20338-DHYD
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Gummy Smile
Keywords: Gingival exposure; Clinical crown length; clinical crown lengthening surgery; Botulinum toxin A; Gummy smile
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Participants were recruited from patients who came for chief complaint of excess gingival display at the Dental Clinic of the Faculty of Odonto-stomatology, University of medicine and Pharmacy at Ho Chi Minh City. The study population included patients aged from eighteen years with an average length of excessive gingival display ≥ of 4 mm when maximum smiling (counted eight teeth, from the 14 to the 24 teeth) and the height of keratinized gingiva ≥ 3 mm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subjects with gummy smile (Experimental): The study procedure consisted of recruitment, pre&post-operative photography, gingivoplasty, BTX-A injection, recall visits, and data collecting.
  Interventions: Procedure: Clinical crown lengthening surgery

INTERVENTIONS:
Procedure: Clinical crown lengthening surgery — * Clinical dental crown lengthening surgery protocol: a clinical crown lengthening surgery was performed.
  * Post-operation protocol Patients were all prescribed antibiotics , anti-inflammation, analgesic, and an antiseptic mouthwash. Patients were instructed for oral hygiene and recalls.
  * Botulinum Toxin A injection One hundred units (U) of botulinum toxin A (BTX-A) were diluted with 2.5ml of sterile saline solution without shaking. 1 mm syringe with a 30-gauge needle was used to get 0.25ml BTX-A for four-point injection, or 0.6ml in case injection of 6 points. Cold compress was applied extraoral 5 mins at injection site before injection.
  After local anesthesia, the doctor administered slowly 2,5 U of diluted BTX-A at each point until white cellulite appeared.
  Patients were recalled two weeks (T2), and two months (T3) after injection.
  Other Names: Botulinum toxin A injection

SUMMARY:
Background: The demand for beauty is increasing in society as everyone is looking for cosmetic improvement, including gummy smile correction.

Object: This study aims to evaluate the efficacy of a combination of a clinical tooth crowns lengthening surgery following by a BTX-A injection in gummy smile treatment upon based on clinical assessment and photography

Method: An uncontrolled longitudinal study was implemented at the Faculty of Odonto-Stomatology (FOS) of the University of Medicine and Pharmacy at Ho Chi Minh City (UMPH), Viet Nam, from August 2020 to May 2021. Twenty patients (19 females and one male) at a mean age of 24 years old who came for gummy smile chief complaint were included in the study. Subjects were operated to lengthen the clinical crown following an additional botulinum toxin A injection two months post-surgery. All the participants answered the smile esthetic satisfactory questions and were photographed at the time before treatment (T0), two months after clinical crown lengthening surgery (T1), two weeks (T2), and two months (T3) follow-up visits after BTX-A injection. The gingival exposure (GE) and clinical crown length (CCL) were measured at each time point for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Gummy smile because of 2 combined etiologies:

  * Short clinical crown of teeth due to the altered passive tooth eruption
  * Hyperactivity of upper lip muscles (lip mobility level > 8mm)

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Gummy smiles due to:

  * Maxillary bone overgrowth (maxillary hypertrophy)
  * Vertical maxillary excess
  * Neuromuscular disorder
  * Gingival hyperplasia due to medicine, supplements, or neuromuscular transmission inhibiting agents
* Systematic diseases that can affect the result of surgical treatment (such as diabetes, heart disease taking blood anticoagulant medicament, blood diseases, immunodeficiency disease etc.)
* Allergy to BTX-A or albumin
* History of taking BTX-A injection in the head-neck area formerly
* Patient with any contraindication of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Gingival exposure | At the time before treatment (T0)
  The outcome is measured in millimeters based on photos of subjects included
Gingival exposure | Two months after clinical crown lengthening surgery (T1)
  The outcome is measured in millimeters based on photos of subjects included
Gingival exposure | Two weeks after Botulinum toxin A injection (T2)
  The outcome is measured in millimeters based on photos of subjects included
Gingival exposure | Two months after Botulinum toxin A injection (T2)
  The outcome is measured in millimeters based on photos of subjects included
Clinical crown length | At the time before treatment (T0)
  The clinical crown length is measured in millimeters using digital caliper and periodontal probe
Clinical crown length | Two months after clinical crown lengthening surgery (T1)
  The clinical crown length is measured in millimeters using digital caliper and periodontal probe
Clinical crown length | Two weeks after Botulinum toxin A injection (T2)
  The clinical crown length is measured in millimeters using digital caliper and periodontal probe
Clinical crown length | Two months after Botulinum toxin A injection (T2)
  The clinical crown length is measured in millimeters using digital caliper and periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Odontostomatology - University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No